CLINICAL TRIAL: NCT03074006
Title: Phase 1/2 Study of Vactosertib (TEW-7197) Monotherapy in Patients With Low or Intermediate Myelodysplastic Syndromes
Brief Title: Dose Escalation and Proof-of-Concept Studies of Vactosertib (TEW-7197) Monotherapy in Patients With MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedPacto, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MP-MDS-01
Record Dates: First submitted 2017-02-27; First posted 2017-03-08 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-06

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- low dose (Experimental)
  Interventions: Drug: TEW-7197
- high dose (Experimental)
  Interventions: Drug: TEW-7197

INTERVENTIONS:
Drug: TEW-7197 — 50mg tablets (doses will be determined through dose-escalation part)

SUMMARY:
This is a prospective, open-label, multicenter, phase 1/2 study of TEW-7197 in patients with low and intermediate risk of myelodysplastic syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible to be included in the study only if they meet all of the following criteria:

1. Subjects who are males or females ≥ 18 years of age.
2. Subjects who are able to give written informed consent.
3. Subjects who have a documented diagnosis of MDS according to WHO criteria.
4. Subjects who have Revised International Prognostic Scoring System (IPSS-R) categories of Very Low, Low- or Intermediate-risk disease. Subjects with cytogenetic failure and ≤ 10% marrow blasts will be eligible.
5. Subjects who meet one of the following hematologic criteria within 8 weeks of registration (according to the IWG criteria) and as documented in prior transfusion logs or weekly hematology evaluations:

   * Symptomatic anemia untransfused with hemoglobin ≤ 9.0 g/dL or with RBC transfusion-dependence (i.e., ≥ 2 units/month) confirmed for a minimum of 8 weeks before randomization.
   * Platelet counts of < 100 x109/L
   * Absolute neutrophil count < 1500
6. Subjects with del(5q) who should have failed or not be a candidate for approved therapy (Lenalidomide) prior to enrolling on this study.
7. Subjects must meet accepted standard criteria for treatment and have failed or not be candidates for standard, accepted treatments.
8. Subjects who have sufficient hepatic function, defined as bilirubin 2 times the upper limit of normal (ULN) and alanine transaminase (ALT) and aspartate transaminase (AST) levels 2.5 times ULN.
9. Subjects who have sufficient renal function, defined as serum creatinine levels 1.5 ULN.
10. Subjects who have a performance status of 2 on the Eastern Cooperative Oncology Group (ECOG) scale (refer to Appendix 2).
11. Subjects who have discontinued all previous therapies for MDS or other investigational therapy for at least 28 days prior to study enrollment and recovered to less than grade 2 toxicity from prior therapy.
12. Subjects who are able to swallow tablets.
13. Subject who are willing and able to comply with scheduled visits, treatment plans, laboratory tests and procedures.
14. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days of the first administration of study drug. For the purpose of this study, female subjects of childbearing potential are defined as all female subjects after puberty unless they are postmenopausal for at least 1 year, or are surgically sterile (hysterectomy or bilateral oophorectomy or tubal ligation).
15. Female subjects of child bearing potential who are willing to avoid the pregnancy during the duration of the study and for 30 days following the last dose of study drug. The effects of TEW-7197 on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
16. Subjects with QTc interval calculated according to Fridericia's formula (QTcF = QT/RR0.33; RR = RR interval) of ≤ 470 ms for males and 450 ms for females on screening electrocardiogram (ECG).
17. Subjects must have ejection fraction more than 50% and no clinically significant valvular dysfunction.
18. Subjects must have discontinued radiotherapy at least 14 days with resolution of any toxicity to Grade 1 or better prior to the start of treatment.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

1. Subjects who have received treatment within the last 28 days with a drug that has not received regulatory approval for any indication at the time of study entry.
2. Subjects who have moderate or severe cardiac disease:
3. Subjects who have the presence of cardiac disease, including a myocardial infarction within 6 months prior to study entry, unstable angina pectoris, New York Heart Association (NYHA) Class III/IV congestive heart failure, or uncontrolled hypertension.
4. Subjects who have documented major electrocardiogram (ECG) abnormalities at the investigator's discretion (for example, symptomatic or sustained atrial or ventricular arrhythmias, second- or third-degree atrioventricular block, bundle branch blocks, ventricular hypertrophy, or recent myocardial infarction).
5. Subjects who have major abnormalities documented by echocardiography with Doppler (for example, moderate or severe heart valve function defect and/or left ventricular ejection fraction (LVEF) <50%, evaluation based on the institutional lower limit of normal).
6. Subjects who have predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress (for example, family history of aneurysms, Marfan-Syndrome, bicuspid aortic valve, evidence of damage to the large vessels of the heart documented by CT scan with contrast).
7. Subjects who have documented iron, B12, folate deficiency as determined by the investigator.
8. Female subjects who are breastfeeding, or intend to breastfeed during the duration of the study and for 30 days following the last dose of study drug.
9. Subjects with any other serious medical condition which in the Investigator's opinion would preclude safe participation in the study.
10. Subjects, in the opinion of the Investigator, who are unsuitable to participate in the study.
11. Subjects with elevated Troponin 1 levels at screening or known to have persistently elevated brain natriuretic peptide (BNP).
12. Subjects with serious pre-existing medical conditions as follows:

    * History of cardiac or aortic surgery,
    * Hypertension that is not controlled by standard medication (to 150/90 mmHg or below),
    * Cirrhosis of the liver, Child-Pugh Stage B or C, or history of liver transplant,
    * Severe diabetes that is not currently controlled,
    * Current or history of interstitial pneumonitis,
    * Presence of aneurisms of the ascending aorta or aortic stress.
13. Subjects with known history of difficulty swallowing, malabsorption or other conditions that may reduce absorption of the product.
14. Subjects with major abnormalities identified by ECG or echocardiogram (ECHO), at the Investigator's discretion.
15. Subjects with active infection with human immunodeficiency virus, hepatitis B virus or hepatitis C virus.
16. Subjects with active infection requiring systemic antibiotic therapy.
17. Subjects who are currently using or planning to use:

Drugs which are exclusively or primarily eliminated by cytochrome P-450 isozyme 3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) for dose escalation phase | 4 weeks
  To define the MTD and determine RP2D
Hematologic improvement (HI) | At 2, 4, 8, 12 and 16 weeks of treatment
  To evaluate the best hematologic improvement (HI) based on IWG 2006 criteria

SECONDARY OUTCOMES:
Hematologic Improvement (HI) | At 2, 4, 8, 12 and 16 weeks of treatment
  To evaluate the duration of HI
Red blood cell transfusion independency | At 2, 4, 8, 12 and 16 weeks of treatment
  To evaluate rate and duration of Red blood cell transfusion independency
Bone marrow response and cytogenetic response | At 2, 4, 8, 12 and 16 weeks of treatment
  To evaluate the frequency of bone marrow response (CP+PR) and cytogenetic response
Time to progression | At 2, 4, 8, 12 and 16 weeks of treatment
  Time to progression to higher risk or acute myeloid leukemia
Relationship between mutations and response | At 2, 4, 8, 12 and 16 weeks of treatment
  To evaluate the relationship between mutations and response
Relationship between various stem and progenitor alterations and response | At 2, 4, 8, 12 and 16 weeks of treatment
  To evaluate the relation ship between various stem and progenitor alterations and response
Quality of life with MDS | At 4, 8, 12 and 16 weeks of treatment
  To evaluate the quality of life parameters experienced by patients with MDS
Biomarker | At 4, 8, 12 and 16 weeks of treatment
  Determine pharmacodynamic markers in bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Sunjin Hwang, MD, Study Chair — MedPacto, Inc.
Locations (3):
- United States (3):
  - Site 03, Tampa, Florida
  - Site 02, Baltimore, Maryland
  - Site 01, The Bronx, New York